CLINICAL TRIAL: NCT00344786
Title: A Phase 1, Dose-Escalation Study of CNF2024 Administered Orally to Patients With B Cell Chronic Lymphocytic Leukemia (CLL)
Brief Title: Phase 1, Dose-Escalation Study of Oral CNF2024(BIIB021) in CLL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNF2024-CLL-05002; 120CL101
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-06

CONDITIONS: B-Cell Chronic Lymphocytic Leukemia
Keywords: CLL; CNF2024; Hsp90 inhibitor
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — 6-chloro-9-(4-methoxy-3,5-dimethylpyridin-2-ylmethyl)-9H-purin-2-ylamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CNF2024 (Experimental)
  Interventions: Drug: CNF2024 (BIIB021)

INTERVENTIONS:
Drug: CNF2024 (BIIB021) — Dose starting at 12.5 mg/d, p.o. as a once-daily dose for 21 days followed by a 1-week rest period.
  Dose escalation will proceed according to the predetermined scheme until the maximum tolerated dose (MTD) is reached due to dose limiting toxicities (DLT) during the first course of treatment.
  Other Names: Single arm trial; no comparator

SUMMARY:
CLL dosing escalating study; daily dosing schedule; PK/PD safety

DETAILED DESCRIPTION:
Phase 1, open-label, accelerated-titration study designed to evaluate the effects of increasing doses of CNF2024 on safety, pharmacokinetics, pharmacodynamic markers, and hematological response

ELIGIBILITY:
Inclusion Criteria:

* Patients with CLL who relapsed following or are intolerant to purine analog -based therapy
* Hemoglobin >=9 gm/dL (may be post-transfusion)
* Total bilirubin <2 X ULN, and ALT and AST <2 x ULN
* Creatinine <=2 X ULN
* Normal plasma cortisol and ACTH concentrations
* ECOG Performance Status <=2
* Anticipated survival >=3 months
* For men and women of child-producing potential, use of effective contraceptive methods during the study and for one month after treatment
* Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and return for the required assessments

Exclusion Criteria:

* Pregnant or nursing women
* Treatment with chemotherapy, monoclonal antibody, or radiotherapy within 28 days before entering the study
* Participation in any investigational drug study within 28 days before CNF2024 administration
* Patients with secondary malignancy requiring active treatment (except hormonal therapy)
* Active symptomatic bacterial, fungal, or viral infection including active HIV or viral (A, B, or C) hepatitis
* Problems with swallowing or malabsorption
* Diarrhea (excess of 2-3 stools/day above normal frequency in the past month)
* Gastrointestinal diseases including gastritis, ulcerative colitis, Crohn's disease, or hemorrhagic coloproctitis
* Major surgery of the stomach or small intestine
* Adrenal dysfunction
* Patients with life- or function-threatening CLL complications (e.g., cord compression, hemolytic crisis, urinary tract obstruction)
* Any illness or condition that in the opinion of the investigator may affect safety of treatment or evaluation of any the study's endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-02; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity (maximum tolerated dose (MTD)) | 4 week periods until MTD is reached
Pharmacokinetics | Dosing period
Pharmacodynamics | Dosing period

SECONDARY OUTCOMES:
To determine clinical and hematological response | Study Duration
To determine the recommended Phase 2 dose | Study duration

CONTACTS AND LOCATIONS:
Overall Officials: Chris Storgard, MD, Study Chair — Biogen
Locations (3):
- United States (3):
  - Research Site, San Diego, California
  - Research site, New York, New York
  - Research site, Houston, Texas